CLINICAL TRIAL: NCT00206674
Title: Phase 3 Randomized, Double-Blind, Placebo Controlled Induction Study of Sargramostim (Leukine®) in Patients With Active Crohn's Disease
Brief Title: Efficacy (Induction of Response/Remission) and Safety Study in Patients With Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 308380; 91405; Novel 4; NCT00185497 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Crohn Disease
Keywords: Morbus Crohn; Sargramostim; Phase III; Placebo Controlled
MeSH Terms: conditions — Crohn Disease | interventions — sargramostim

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Sargramostim (Leukine)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sargramostim (Leukine) — 6µg/kg SARGRAMOSTIM subcutaneous daily for 8 weeks
  Other Names: BAY86-5326
  Arms: Arm 1
Drug: Placebo — Sterile liquid solution, inactive excipient only subcutaneous daily for 8 weeks
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate if Leukine can induce clinical response or remission in patients with Crohn's disease.

DETAILED DESCRIPTION:
On 29 May 2009, Bayer began transitioning the sponsorship of this trial to Genzyme. NOTE: This study was originally posted by sponsor Berlex, Inc. Berlex, Inc. was renamed to Bayer HealthCare, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Stable but active Crohn's disease at the time of screening
* Must be able to self-inject or have another person who can help with the injection

Exclusion Criteria:

* Not have a colostomy or ileostomy
* Not be taking prohibited medications as defined in the protocol
* Not have had GI surgery or a bowel obstruction in the last 6 months or planned surgery for the next months
* Not have ever taken this drug or drugs of similar type in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2004-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Induction of clinical response and/or remission as defined by decrease in CDAI score | After 8 weeks of treatment

SECONDARY OUTCOMES:
Time and duration to response/remission | During the 8 weeks of treatment
QoL (different methods) | During the whole study
Safety Profile ( Adverse Event, Serious Adverse Event collection, laboratories especially AB test etc.) | About 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (59):
- Buenos Aires, Buenos Aires F.D., Argentina
- Australia (14):
  - Garran, Australian Capital Territory
  - Concord, New South Wales
  - New Lambton Heights, New South Wales
  - Sydney, New South Wales
  - Brisbane, Queensland
  - Adelaide, South Australia
  - Launceston, Tasmania
  - Ballarat, Victoria
  - Frankston, Victoria
  - Melbourne, Victoria
  - Parkville, Victoria
  - Prahran, Victoria
  - Fremantle, Western Australia
  - Penrith
- Brazil (5):
  - Salvador, Estado de Bahia
  - Curitiba, Paraná
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Canada (12):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
- New Zealand (3):
  - Milford, Auckland
  - Christchurch
  - Hamilton
- Russia (6):
  - Lipetsk, Russia
  - Moskva, Russia
  - Samara, Russia
  - Moscow
  - Moskva
  - Volgograd
- Switzerland (3):
  - Basel, Basel
  - Bern, Canton of Bern
  - Lausanne, Canton of Vaud
- Ukraine (5):
  - Donetsk
  - Kharkiv
  - Kiev
  - Lviv
  - Vinnitsa
- United Kingdom (10):
  - Bristol, Avon
  - London, Greater London
  - Salford, Greater Manchester
  - Edinburgh, Lothian
  - Liverpool, Merseyside
  - Harrow, Middlesex
  - Cardiff, South Glamorgan
  - Newcastle upon Tyne, Tyne and Wear
  - London
  - Sheffield